CLINICAL TRIAL: NCT06394479
Title: Evaluation of the Long-term Outcome After Bariatric Surgery in Patients With Type 1 Diabetes Mellitus
Brief Title: Long-term Results After Bariatric Surgery in Type 1 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: Sana Klinikum Offenbach (Other)
Collaborators: SRH Wald-Klinikum Gera GmbH (Other); Wuerzburg University Hospital (Other); Kuwait University (Other); Cleveland Clinic Florida (Other)
Responsible Party: Principal Investigator, Christine Stier, Study coordinator, Sana Klinikum Offenbach
Other Study IDs: FF120/2015
Record Dates: First submitted 2019-12-06; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Bariatric Surgery Status in T1D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Outcome after bariatric surgery in patient with T1D — Retrospective evaluation of clinical data
  Other Names: Metabolic changes after bariatric surgery in T1D

SUMMARY:
There is a lack of long-term data on the impact of bariatric surgery in type 1 diabetes (T1D). The aim of this study is to gain long-term outcome data on the effects of bariatric surgery in obese patients with T1D.

DETAILED DESCRIPTION:
This study aims to evaluate long-term data on the effect of bariatric surgery in T1D regarding weight lost, insulin-requirement, and quality of life.

Inclusion criteria are patients who underwent bariatric surgery (Sleeve, One anastomosis gastric bypass, Roux en Y Gastric Bypass) and the presence of T1D prior to surgery. Labor parameters include verification of T1D antibodies, and level of C-peptide. Exclusion criteria is T2D.

In order to obtain a sufficient number of patients for the evaluation, several sites are involved in the acquisition of these specific data.

ELIGIBILITY:
Inclusion Criteria:

* T1D-specific antibodies
* C-peptide level
* status after bariatric surgery

Exclusion Criteria:

* T2D
* patients without T1D
* patients with T1d without bariatric surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with T1D, who underwent bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Post-surgical impact on body weight | 1 year
  Body weight in kgpost-surgical A1c course

SECONDARY OUTCOMES:
Post-surgical impact on metabolic changes | 1 year
  insulin-requirement in I.U.
Post-surgical impact on body weight and metabolic changes | 1 year
  insulin-requirement per kg/BW

CONTACTS AND LOCATIONS:
Overall Officials: Christine Stier, MD, Study Director — Sana Klinikum Offenbach
Locations (1):
- Sana obesity center, Remscheid, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirwan JP, Aminian A, Kashyap SR, Burguera B, Brethauer SA, Schauer PR. Bariatric Surgery in Obese Patients With Type 1 Diabetes. Diabetes Care. 2016 Jun;39(6):941-8. doi: 10.2337/dc15-2732. PMID 27222552
- [Background] Chillaron JJ, Flores Le-Roux JA, Benaiges D, Pedro-Botet J. Type 1 diabetes, metabolic syndrome and cardiovascular risk. Metabolism. 2014 Feb;63(2):181-7. doi: 10.1016/j.metabol.2013.10.002. Epub 2013 Oct 24. PMID 24274980
- [Background] Fourlanos S, Narendran P, Byrnes GB, Colman PG, Harrison LC. Insulin resistance is a risk factor for progression to type 1 diabetes. Diabetologia. 2004 Oct;47(10):1661-7. doi: 10.1007/s00125-004-1507-3. Epub 2004 Oct 6. PMID 15480539
- [Background] Lannoo M, Dillemans B, Van Nieuwenhove Y, Fieuws S, Mathieu C, Gillard P, D'Hoore A, Van Der Schueren B. Bariatric surgery induces weight loss but does not improve glycemic control in patients with type 1 diabetes. Diabetes Care. 2014 Aug;37(8):e173-4. doi: 10.2337/dc14-0583. No abstract available. PMID 25061146
- [Background] Polsky S, Ellis SL. Obesity, insulin resistance, and type 1 diabetes mellitus. Curr Opin Endocrinol Diabetes Obes. 2015 Aug;22(4):277-82. doi: 10.1097/MED.0000000000000170. PMID 26087341
- [Background] Chillaron JJ, Benaiges D, Mane L, Pedro-Botet J, Flores Le-Roux JA. Obesity and type 1 diabetes mellitus management. Minerva Endocrinol. 2015 Mar;40(1):53-60. Epub 2014 Nov 21. PMID 25413942
- [Background] Corbin KD, Driscoll KA, Pratley RE, Smith SR, Maahs DM, Mayer-Davis EJ; Advancing Care for Type 1 Diabetes and Obesity Network (ACT1ON). Obesity in Type 1 Diabetes: Pathophysiology, Clinical Impact, and Mechanisms. Endocr Rev. 2018 Oct 1;39(5):629-663. doi: 10.1210/er.2017-00191. PMID 30060120
- [Background] Mahawar KK, De Alwis N, Carr WR, Jennings N, Schroeder N, Small PK. Bariatric Surgery in Type 1 Diabetes Mellitus: A Systematic Review. Obes Surg. 2016 Jan;26(1):196-204. doi: 10.1007/s11695-015-1924-z. PMID 26452482
- [Background] Ashrafian H, Harling L, Toma T, Athanasiou C, Nikiteas N, Efthimiou E, Darzi A, Athanasiou T. Type 1 Diabetes Mellitus and Bariatric Surgery: A Systematic Review and Meta-Analysis. Obes Surg. 2016 Aug;26(8):1697-704. doi: 10.1007/s11695-015-1999-6. PMID 26694210
- [Background] Mottalib A, Kasetty M, Mar JY, Elseaidy T, Ashrafzadeh S, Hamdy O. Weight Management in Patients with Type 1 Diabetes and Obesity. Curr Diab Rep. 2017 Aug 23;17(10):92. doi: 10.1007/s11892-017-0918-8. PMID 28836234
- [Background] Hussain A. The effect of metabolic surgery on type 1 diabetes: meta-analysis. Arch Endocrinol Metab. 2018 Apr 5;62(2):172-178. doi: 10.20945/2359-3997000000021. Print 2018 Mar-Apr. PMID 29641734
- [Background] Akcay MN, Karadeniz E, Ahiskalioglu A. Bariatric/Metabolic Surgery in Type 1 and Type 2 Diabetes Mellitus. Eurasian J Med. 2019 Feb;51(1):85-89. doi: 10.5152/eurasianjmed.2018.18298. PMID 30911264
- [Background] Landau Z, Kowen-Sandbank G, Jakubowicz D, Raziel A, Sakran N, Zaslavsky-Paltiel I, Lerner-Geva L, Pinhas-Hamiel O. Bariatric surgery in patients with type 1 diabetes: special considerations are warranted. Ther Adv Endocrinol Metab. 2019 Jan 30;10:2042018818822207. doi: 10.1177/2042018818822207. eCollection 2019. PMID 30728940